CLINICAL TRIAL: NCT02477683
Title: Pilot Evaluation of the FilmArray® Febrile Infant (FI) Panel
Status: Completed | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BFDxFIPilot
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Acute Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and Whole Blood

SUMMARY:
The purpose of this study is to collect data to support decisions made by BioFire regarding assay development, panel composition, and intended use for the final FilmArray FI reagent pouch. The study will utilize whole blood and/or plasma obtained from pediatric patients under 3 years of age that present with acute fever.

ELIGIBILITY:
Inclusion Criteria:

* under age of 3
* has fever with no obvious focal infection
* written informed parental permission

Exclusion Criteria:

* parent/legal guardian unable to provide permission
* participation determined by a physician to be detrimental to patient health

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients under the age of 3 with acute fever.
Sampling Method: Non-Probability Sample
Enrollment: 1514 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Utility of multiplexed testing for pathogens in pediatric patients with acute fever | 15 months

SECONDARY OUTCOMES:
Epidemiology of pathogens in pediatric patients with acute fever | 15 Months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medecine, Indianapolis, Indiana
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah